CLINICAL TRIAL: NCT00437138
Title: The Effects of Air Pollution on Vascular and Endogenous Fibrinolytic Function in Patients With Coronary Heart Disease
Brief Title: Controlled Exposures to Air Pollution in Patients With Coronary Heart Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Umeå University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: RG/05/003 DISARM 2
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2007-02-19 (Estimated); Status verified 2007-02

CONDITIONS: Coronary Heart Disease
Keywords: Air pollution; Myocardial ischemia; Endothelium; Fibrinolysis; Pathophysiology; Diesel exhaust
MeSH Terms: conditions — Coronary Disease; Myocardial Ischemia

INTERVENTIONS:
Behavioral: Exposure to dilute diesel exhaust (300µg/m3) or filtered air

SUMMARY:
Air pollution is a major cause of cardiovascular morbidity and mortality. The components of air pollution responsible and the mechanisms through which they might mediate these harmful effects remain only partially understood. We hypothesise that these adverse effects are mediated by combustion derived air pollutants and that even a brief exposure will effect heart and blood vessel function. We assess the effect of dilute diesel exhaust inhalation at levels encountered in urban road traffic on heart and blood vessel function in patients with stable coronary heart disease.

DETAILED DESCRIPTION:
Observational studies suggest that exposure to air pollution may worsen symptoms of angina and trigger acute myocardial infarction. These findings are limited by imprecision in the measurement of pollution exposure, the effect of potential confounding environmental and social factors, and the lack of mechanistic data. Controlled exposures of air pollutants can help to address these shortcomings by providing a precisely defined exposure in a regulated environment that facilitates investigation with validated biomarkers and surrogate measures of cardiovascular health. Using a carefully characterised exposure system, we have previously shown in healthy volunteers that exposure to dilute diesel exhaust causes lung inflammation, depletion of airway antioxidant defences, and impairment of vascular and fibrinolytic function. To date, there have been no controlled exposures in patients with coronary heart disease: an important population who may be particularly susceptible to the adverse cardiovascular effects of air pollution.

In a double blind randomized cross-over study, 20 patients with prior myocardial infarction will be exposed to dilute diesel exhaust (300µg/m3) or filtered air during periods of rest and moderate exercise in a controlled exposure facility. During the exposure, myocardial ischemia will be quantified by ST-segment analysis using continuous 12-lead electrocardiography. Six hours following exposure, vascular vasomotor and fibrinolytic function will be assessed by means of intra-arterial agonist infusions.

ELIGIBILITY:
Inclusion Criteria:

* Previous myocardial infarction (>6 months previously) treated by primary angioplasty and stenting
* On standard secondary preventative therapy

Exclusion Criteria:

* Angina pectoris (Canadian Cardiovascular Society grade ≥2)
* History of arrhythmia
* Diabetes mellitus
* Uncontrolled hypertension
* Renal or hepatic failure
* Unstable coronary disease (acute coronary syndrome or unstable symptoms within 3 months)
* Occupational exposure to air pollution
* Current smokers
* Asthma
* Inter-current illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-04; Study Completion 2006-06

PRIMARY OUTCOMES:
Exercise induced myocardial ischemia
Vascular vasomotor function
Endogenous fibrinolytic function

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, MD, Principal Investigator — University of Edinburgh; Thomas Sandstrom, MD, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Umeå, Västerbotten County, Sweden

REFERENCES:
- [Derived] Langrish JP, Watts SJ, Hunter AJ, Shah AS, Bosson JA, Unosson J, Barath S, Lundback M, Cassee FR, Donaldson K, Sandstrom T, Blomberg A, Newby DE, Mills NL. Controlled exposures to air pollutants and risk of cardiac arrhythmia. Environ Health Perspect. 2014 Jul;122(7):747-53. doi: 10.1289/ehp.1307337. Epub 2014 Mar 25. PMID 24667535
- [Derived] Mills NL, Tornqvist H, Gonzalez MC, Vink E, Robinson SD, Soderberg S, Boon NA, Donaldson K, Sandstrom T, Blomberg A, Newby DE. Ischemic and thrombotic effects of dilute diesel-exhaust inhalation in men with coronary heart disease. N Engl J Med. 2007 Sep 13;357(11):1075-82. doi: 10.1056/NEJMoa066314. PMID 17855668
- See also: Centre for Cardiovascular Science, Edinburgh — http://www.cvs.med.ed.ac.uk/
- See also: British Heart Foundation — http://www.bhf.org.uk/